CLINICAL TRIAL: NCT04225559
Title: Analysis of Gastrointestinal Symptoms of Outpatients With Functional Gastrointestinal Diseases（FGIDs） in Grade-A Tertiary Hospitals in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: XL018
Record Dates: First submitted 2019-12-29; First posted 2020-01-13 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2019-12

CONDITIONS: To Analyze TCM Syndrome and Symptoms of FGIDs Patients

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To analyze the classification characteristics of gastrointestinal symptoms, the quality of life, the degree of anxiety and depression, and the satisfaction with the treatment of Chinese medicine in patients with FGIDs in Chinese Grade-A Tertiary Hospitals.

The characteristics of TCM（Traditional Chinese Medicine） syndromes and symptoms of the above-mentioned FGIDs will be analyzed, and the characteristics of TCM syndromes of FGIDs and their possible relationship with FGIDs subtypes will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms has appeared for at least 3 months;
2. No organic disease and gastrointestinal alarm symptoms, which meet the diagnostic criteria of FGIDs;
3. Sign informed consent and be able to read and understand the questionnaire.

Exclusion Criteria:

1. A history of organic gastrointestinal diseases;
2. Alarm symptoms of digestive tract (such as melena, weight loss, fever, abdominal mass, ascites, anemia, family history of gastrointestinal tumors, etc.)
3. Have a history of mental diseases;
4. Unable to read and understand the questionnaire.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients in Chinese Grade-A tertiary hospitals who has been diagnosed FGIDs
Sampling Method: Probability Sample
Enrollment: 4632 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Rome IV functional gastrointestinal disease diagnosis questionnaire | baseline
  Fill in only at the time of the patient's consultation, to assess the patient's current situation.Investigation of patients with functional gastrointestinal symptoms according to Rome IV diagnostic criteria.Determine the type of disease based on the questionnaire.

SECONDARY OUTCOMES:
PHQ-15 Scale | baseline
  Fill in only at the time of the patient's consultation, to assess the patient's current situation.Score evaluation from of physical symptoms in patients with functional gastrointestinal disorders from 15 aspects. 0-4 points: very mild， 5-9 points: mild ，10-14 points: moderate，15-30 points: severe.
SF-36 Scale | baseline
  Fill in only at the time of the patient's consultation, to assess the patient's current situation.Score evaluation from 8 aspects: physical function, role-physical, pain, global health status, vitality，social function,role-emotional， mental health.Use score changes to assess improvement in all areas of the patient. Maximum score is147.The higher the score, the better the status in all aspects.
Hospital Anxiety and Depression Scale (HADS) | baseline
  Fill in only at the time of the patient's consultation, to assess the patient's current situation.Scoring to determine if a patient has symptoms of anxiety and depression：(0-7: asymptomatic， 8-10: suspicious symptoms， 11-21: there must be symptoms).

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - Xiyuan hospital, Beijing, Beijing Municipality
  - Beijing Hospital of Traditional Chinese Medicine, Capital Medical University, Dongcheng, Beijing Municipality
  - Guang'anmen Hospital,China Academy of Chinese Medical Science, Xicheng, Beijing Municipality
  - The Second Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Liuzhou Traditional Chinese Medical Hospital, Liuchow, Guangxi
  - The First Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, Henan
  - Wuhan Hospital Of Traditional Chinese And Western Medicine(WUHAN No.1 HOSPITAL), Wuhan, Hubei
  - Inner Mongolia Autonomous Region Hospital Chinese Medicne, Hohhot, Inner Mongolia
  - Jiangsu Provincial Hospital of Chinese Medicine, Nanjing, Jiangsu
  - The Affiliated Hospital of Liaoning University of Traditional Chinese Medicine,, Shenyang, Liaoning
  - The Affiliated Hospital of Shaanxi, University of Chinese Medicine,, Xianyang, Shaanxi
  - Institute of Digestive Diseases, Longhua Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Shanxi Provincial Hospital Of Traditional Chinese Medicine, Taiyuan, Shanxi
  - First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - Hong Kong Chinese Medicine Clinical Study Centre, Hong Kong
  - School of Chinese Medicine,Hong Kong Baptist University, Hong Kong